CLINICAL TRIAL: NCT06985914
Title: Retrospective Study of CT Scan Indications in Adult Emergency Departments: Are They Justified and Aligned With Official Guidelines
Brief Title: Retrospective Study of CT Scan Indications in Adult Emergency Departments
Acronym: IMA-URG
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Intercommunal de Toulon La Seyne sur Mer (Other)
Responsible Party: Sponsor
Other Study IDs: 2025-CHITS-009
Record Dates: First submitted 2025-05-15; First posted 2025-05-22 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: CT Scan
Keywords: CT Scan; Recommandations; Emergency; patent management
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CT scan patient cohort: Adult patient who received a CT scan in the emergency department in 2024
  Interventions: Procedure: CT scan

INTERVENTIONS:
Procedure: CT scan — CT scan in the emergency department

SUMMARY:
The use of CT scans has significantly improved the diagnosis of various pathologies in emergency departments. However, it is also associated with several drawbacks, including high costs and a proven carcinogenic risk to patients, depending on the dose of radiation received. Furthermore, the ecological impact of this imaging modality should not be overlooked, as each CT scan generates approximately 2 kg of CO₂, contributing to global warming. These concerns underscore the importance of ensuring that CT scans are performed only when clinically justified.

This context motivated our study: a retrospective, descriptive analysis conducted in the emergency department of Sainte Musse Hospital over a 28-day period in 2024. The selected days are distributed to reflect an equivalent representation of weekdays, weekends, and public holidays, as well as seasonal variations.

Our primary objective is to calculate the proportion of CT scans that were appropriately justified. The investigators will assess three key metrics:

* The rate of CT scans justified based on official clinical guidelines.
* The rate of CT scans justified by a change in patient management.
* The rate of CT scans performed at the request of a specialist consulted during the emergency department visit.

The ultimate aim of our study is to evaluate the extent of potential overuse of CT scans in the emergency setting and, if applicable, to raise awareness among emergency physicians regarding the importance of balancing clinical benefit against potential risks for the patient.

DETAILED DESCRIPTION:
CT scans are widely used in modern emergency departments, facilitating the diagnosis of both urgent and non-urgent conditions. However, a noticeable increase in the use of imaging-particularly CT scans-has been observed in recent years. This trend can be attributed to several factors, including technological advancements that have made imaging more accessible, as well as a rising number of patients presenting to emergency departments.

Nevertheless, studies have raised concerns about the appropriateness of this increase. Notably, Keith E. Kocher et al. reported that between 1996 and 2007, the number of emergency department visits in a U.S. hospital increased by 30%, while the number of CT scans performed rose by an astonishing 330% over the same period. This disproportionate rise raises questions about the justification of many of these examinations, especially considering the potential consequences-ranging from increased healthcare costs and radiation exposure to environmental impact.

Imaging examinations such as CT scans are associated with significant costs and expose patients to ionizing radiation. It has been demonstrated that CT-related radiation is linked to an increased risk of cancer, particularly with high or cumulative doses, thereby posing a public health concern. In addition, the environmental impact of CT imaging should not be overlooked: each scan generates approximately 2 kg of CO₂, contributing to global warming. These concerns highlight the importance of using CT scans judiciously and minimizing unjustified imaging whenever possible, in order to limit both medical and ecological consequences.

At the international level, several studies have highlighted significant variability in the rate of unjustified CT scans. For example, Heljä Oikarinen et al. (2009) reported that in a Swedish hospital radiology department, 77% of lumbar spine CT scans, 36% of brain CT scans, and 37% of abdominal CT scans were unjustified in patients under the age of 35. More recently, Andreas Sakkas et al. (2023) found that 37.8% of brain CT scans performed for head trauma in a German maxillofacial surgery department were unjustified. In contrast, Aleksandra Sobiecka et al. (2019) reported a much lower rate-only 6.54% of CT and MRI scans were deemed unjustified-across two radiology departments in Poland.

These divergent findings from country to country underscore the complexity of assessing imaging appropriateness and highlight the need for local evaluations. Given the public health implications in France-including healthcare costs and radiation exposure-as well as the global environmental impact of medical imaging, the investigators have undertaken a retrospective observational study in the adult emergency department of Hôpital Sainte Musse. The objective is to assess the justification of CT scans prescribed in this setting. More specifically, the investigators aim to calculate the proportion of CT scans that are justified either by adherence to official clinical guidelines or by a subsequent change in patient management resulting from the imaging findings.

Keith E. Kocher et al. have shown that the overuse of imaging tests in emergency departments may be associated with a reduction in hospital admissions. In light of this, the investigators have defined secondary objectives in our study: to assess the proportion of CT scans justified by adherence to official clinical guidelines and the proportion justified by a change in patient management. For the latter, the investigators will characterize the nature of the management change, such as the initiation of appropriate treatment or a modification in patient disposition (e.g., discharge home, arrangement of outpatient follow-up, hospital admission, and transfer to another facility, or referral to the operating room).

Additionally, the investigators have observed that a portion of CT scans performed in the emergency department are ordered at the request of specialists consulted during the patient's visit. These specialists may prefer to request imaging through the emergency department due to limited access to imaging resources in inpatient units, thereby avoiding delays in patient care. Consequently, they will also calculate the rate of justified CT scans ordered by specialists but performed within the emergency department.

ELIGIBILITY:
Inclusion Criteria:

* Adults (> 18 years)
* CT scans performed in emergencies in 2024 at Hôpital Ste Musse -

Exclusion Criteria:

1. CT scans performed outside the emergency department
2. Patients managed through the neurovascular pathway
3. Patients under protective supervision (e.g., guardianship or legal protection)
4. Patients who refuse to participate in the research -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (≥ 18 years) who received a CT scan during a visit to the emergency department of Hôpital Ste Musse during the period 01/01/2024 to 31/12/2024.
Sampling Method: Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
rate of justified CT scans performed in adult emergency settings | up to 12 months
  The rate of justified emergency CT scans is defined as the proportion of CT scans performed in the adult emergency department that are either compliant with the recommendations of the Société Française de Réanimation (SFR) and/or have had a documented impact on patient management, relative to the total number of CT scans performed during a randomly selected sample of 28 days over a one-year period.

SECONDARY OUTCOMES:
Evaluate the rate of justified emergency CT scans according to official recommendations. | up to 12 months
  The rate of justified emergency CT scans is defined as the proportion of CT scans performed in the emergency department that are assessed as compliant with official recommendations, relative to the total number of CT scans performed in the emergency department.
Evaluate the rate of emergency CT scans assessed as having had an impact on patient management | up to 12 months
  The rate of justified emergency CT scans is defined as the proportion of CT scans performed in the emergency department that are assessed as having had an impact on patient management-whether therapeutic and/or related to patient referral-relative to the total number of CT scans performed in the emergency department.
evaluate the rate of emergency CT scans, requested by specialists | up to 12 months
  The percentage of CT scans requested by specialists-categorized by specialty-that are justified, either by conformity with official recommendations and/or by having had a documented impact on patient management.

CONTACTS AND LOCATIONS:
Overall Officials: Tiziana Platino, MD, Study Director — CHITS
Locations (1):
- CHITS, Toulon, VAR, France